CLINICAL TRIAL: NCT00707057
Title: Ibuprofen 600 mg Extended-Release (ER) Multiple-Dose Dental Pain Study
Brief Title: Ibuprofen Extended-Release Dental Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SCOLR Pharma, Inc. (Industry)
Collaborators: AAIPharma (Industry); Jean Brown Research (Other)
Responsible Party: Stephen Turner, President & CEO, SCOLR Pharma, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCO-0001
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Pain; Post-Operative Pain; Third Molar Extraction
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen 600 mg ER group (Experimental): One-hundred and sixty subjects will be randomly assigned to the Ibuprofen 600 mg ER treatment group based on gender and baseline pain intensity, as rated on an 11-point numerical rating scale (PI-NRS; 5-7 moderate pain, or 8-10, severe pain).
  Interventions: Drug: Ibuprofen 600 mg Extended-Release Tablets
- Placebo group (Placebo Comparator): Eighty subjects will be randomly assigned to the Placebo treatment group based on gender and baseline pain intensity, as rated on an 11-point numerical rating scale (PI-NRS; 5-7 moderate pain, or 8-10, severe pain).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 600 mg Extended-Release Tablets — Ibuprofen 600 mg Extended-Release Tablet: One 600 mg tablet taken orally every 12 hours or twice daily (BID). Each dose was administered with at least 6 ounces of water. Dose 1 was administered at hour 0, Dose 2 was administered at hour 12, Dose 3 was administered at hour 24 and Dose 4 was administered at hour 36.
  Other Names: Ibuprofen 600 mg ER
  Arms: Ibuprofen 600 mg ER group
Drug: Placebo — Placebo: One matching placebo tablet was taken orally every 12 hours or twice daily (BID). Each dose was administered with at least 6 ounces of water. Dose 1 was administered at hour 0, Dose 2 was administered at hour 12, Dose 3 was administered at hour 24 and Dose 4 was administered at hour 36.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of multiple doses of Ibuprofen 600 mg Extended-Release Tablets in a study of dental pain following extraction of third molar teeth.

DETAILED DESCRIPTION:
This is a single-center, multiple-dose, randomized, placebo-controlled, double-blinded, parallel group trial to evaluate the efficacy and safety of multiple doses of Ibuprofen 600 mg Extended-Release Tablets in a study of dental pain following extraction of third molar teeth. The surgery will consist of surgical extraction of 1-2 impacted third molars, of which one must be a mandibular impaction that is partially impacted in either tissue or bone. Subjects will be stratified according to baseline pain intensity, as rated on an 11-point pain intensity numerical rating scale (PI-NRS)and gender.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16 to 45 years of age;
* Outpatients scheduled to undergo surgical extraction of 1-2 impacted third molar(s), one of which must be a mandibular impaction that is partially impacted in either tissue or bone;
* At least a score of 5 on the 11-point pain intensity numerical rating scale (PI-NRS) at baseline;
* Use of only the following preoperative medication(s) / anesthetic(s): short-acting local anesthetic (e.g., mepivacaine or lidocaine) with or without vasoconstrictor and/or nitrous oxide;
* Reliable, cooperative, and adequate intelligence to record the requested information on the analgesic questionnaire form;
* Subjects (or the parent or legal guardian of subjects under the age of 18 years) are required to read, comprehend, and sign the informed consent. Subjects requiring a parent or legal guardian to sign the informed consent will be required to sign an assent;
* Examined by the attending dentist or physician and medically cleared to participate in the study; and,
* In general good health and have no contraindications to any of the study meds.

Exclusion Criteria:

* Presence of a serious medical condition (e.g., poorly controlled hypertension, poorly controlled diabetes, significantly impaired cardiac, renal or hepatic function, hyper- or hypothyroidism);
* Use of a prescription or nonprescription drug with which the administration of ibuprofen, celecoxib, any other non-steroidal anti-inflammatory drug (NSAID), or acetaminophen, is contraindicated;
* Acute local infection at the time of surgery that could confound the post-surgical evaluation;
* Females who are pregnant, lactating, of child-bearing potential, or postmenopausal for less than 2 years and not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a urine-based pregnancy test;
* Presence or history (within 2 years of enrollment) of bleeding disorder(s) or peptic ulcer disease;
* Presence or history (within the past year) of alcoholism or substance abuse. Subjects who are taking CNS or other psychotropic drugs (including St. John's Wort, or any other nutritional supplement known to have psychotropic effects) may be enrolled if they have been on stable doses of medication for at least 2 months, will maintain this dose throughout the study, and their condition is judged by the Principal Investigator to be well-controlled;
* Habituation to analgesic drugs (i.e., routine use of oral analgesics 5 or more times per week);
* History of allergic reaction (eg, asthma, rhinitis, swelling, shock, or hives) to ibuprofen, naproxen, aspirin, celecoxib, any other NSAID, or acetaminophen;
* Prior use of any type of analgesic or NSAID 5 half-lives of that drug or less before taking the first dose of study medication, except for pre-anesthetic medication and anesthesia for the procedure;
* Ingestion of any caffeine-containing beverages, chocolate, or alcohol 4 hours or less before taking the first dose of study medication;
* Has taken an investigational product within the past 30 days;
* Has previously been entered into this study; and,
* The subject is a member of the study site staff either directly involved with the study, an employee of the Sponsor, or a relative of study site personnel directly involved with the study or Sponsor.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 256 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Christensen, D.D.S., Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date First Subject Enrolled: 24 June 2008 Date Last Subject Enrolled: 11 October 2008 All subjects were to receive 4 doses of study drug or placebo at 12-hour intervals. Of the 12 subjects who prematurely discontinued study drug, 6 subjects received 1 dose of study drug, 2 subjects received 2 doses, and 4 subjects received 3 doses.
Groups:
- Ibuprofen 600mg ER: Participants received 600 mg 12-hour extended-release tablets twice daily (BID).
- Placebo: Participants received placebo tablet twice daily (BID)
Period: Overall Study
Arm/Group | Ibuprofen 600mg ER | Placebo
Started | 169 | 87
Completed | 161 | 83
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Dosed incorrectly | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen 600mg ER | Placebo | Total
Number analyzed (Participants) | 169 | 87 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 35 | 99
  Between 18 and 65 years | 105 | 52 | 157
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.9 (3.22) | 18.8 (3.25) | 18.9 (3.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 47 | 142
  Male | 74 | 40 | 114
Region of Enrollment [Number; unit: participants]
  United States | 169 | 87 | 256

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Efficacy, as Measured by the Sum of Pain Intensity Differences (SPID) Scale
Description: Analgesic efficacy for the 8-12 hour measurement interval after dose 1 using Sum of Pain Intensity Differences (SPID).
  An 11-point Pain Intensity Numerical Rating Scale (PI-NRS) was used to record pain intensity at baseline and 8, 9, 10, 11, 12 hours after dose 1. The scale went from 0 (no pain) to 10 (Worst possible pain). The outcome measure is based a mean of the sum of each of the five time points evaluated. The total time scale ranges from 0 to 50. Subjects were asked to select the number that best describes how much pain they had at the time of observation.
Time Frame: from baseline to 12 hours after dose 1
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale | 14.80 (16.331) [0.65 to 0.78] | 0.40 (11.933) [0.23 to 0.43]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; The null versus alternative hypothesis regarding the analgesic efficacy using the SPID 8-12 was compared between the 2 treatment groups using an analysis of covariance (ANCOVA)model with each subject's outcome being his/her SPID 8-12 as the dependent variable in the ANCOVA model with terms for gender, treatment, and baseline pain score categories (stratified as ≤7 and >7); Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Primary Outcome: Durability of Effect as Measured by the Number of Subjects Achieving Meaningful Improvement in Pain Intensity Difference (PID) From Baseline at All Three Assessment Periods of 24, 36, and 48 Hours
Description: Response rate measured the durability of effect and was measured by the number of subjects achieving a reduction of at least 2 points (greater than or equal to 20%) from baseline on the 11-point Pain Intensity Numerical Rating Scale (PI-NRS) at all 3 assessment periods of 24, 36 and 48 hours. The scale went from 0 (no pain) to 10 (Worst possible pain). Subjects were asked to select the number that best describes how much pain they had at the time of observation.
Time Frame: 24, 36, and 48 hours
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
participants | 123 | 47
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; The null versus alternative hypothesis regarding the durability of analgesic efficacy using the PID scores at 24, 36, and 48 hours.An individual subject was to achieve the 2-point reduction at all 3 terminal time points in order to be defined as responder; Test type: Superiority or Other; p < 0.0017, ANCOVA

3. Secondary Outcome: Time to Confirmed "First Perceptible" Relief
Description: When the subject was administered study medication at Time 0, the Study Coordinator started 2 stopwatches. In an effort to determine the exact moment that the subject began to obtain noticeable pain relief, the subject was instructed to stop the stopwatch when "initial" relief was observed and again when "meaningful" relief was achieved. Time to confirmed first perceptible relief was defined as the time to first perceptible relief, provided that the subject also later stopped the second stopwatch indicating meaningful relief. The assigned censored time for "No Pain Relief" is 240 minutes.
Time Frame: Within 4 hours post Dose 1
Population: Intention to treat (ITT)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Minutes | 42.00 [4 to 81] | 240 [240 to 240]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Time to confirmed first perceptible relief was defined as the time to first perceptible relief, provided that the subject also stopped the second stopwatch indicating meaningful relief. For those who failed to achieve confirmed first perceptible and/or meaningful relief, a censored time was assigned; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Time to Confirmed "Meaningful" Relief
Description: When the subject was administered study medication at Time 0, the Study Coordinator started 2 stopwatches. To determine the exact moment that the subject began to notice pain relief, the subject was instructed to stop the stopwatch when "initial" relief was observed and again when "meaningful" relief was achieved. Time to confirmed "meaningful" relief was achieved if both stopwatches were stopped within the 4 hour observation period, when both "initial" and "meaningful" relief were observed. Meaningful relief is a subjective definition, based on each subjects determination of pain.
Time Frame: Within 4 hours post Dose 1
Population: Intention to treat (ITT)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Minutes | 108 [18 to 240] | 240 [240 to 240]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage (%) of Subjects With Confirmed First Perceptible Relief Within 1 Hour of Dose 1
Description: Percentage (percentage of total) of subjects with "first perceptible" relief within 1 hour of Dose 1. The assigned censored time for "No Pain Relief" was 240 minutes.
Time Frame: Within 1 hour of Dose 1
Population: Intention to treat (ITT)
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Percent of participants | 62 [54 to 69] | 12 [5 to 18]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Subjects Achieving "Meaningful" Relief as Indicated by the Time Recorded on the Second Stopwatch Following "First Perceptible" Relief
Description: Percentage(%) of subjects with confirmed first perceptible relief and meaningful relief after dose 1. Subjects that achieved both "first perceptible" relief and "meaningful" relief within the time allotted. The assigned censored time for "No Pain Relief" is 240 minutes. Meaningful relief is a subjective definition, based on each subject's determination of pain
Time Frame: Within 4 hours post Dose 1
Population: Intention to treat (ITT)
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Percent of participants | 69 [62 to 76] | 17 [9 to 25]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Ibuprofen 600mg ER vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Estimated Confidence Interval: 95%Method: Cochran-Mantel-Haenszel

7. Secondary Outcome: Analgesic Efficacy for the 0-12, 0-4, 4-8, and 4-12 Hour Dosing Intervals After Dose 1 Using Total Pain Relief (TOTPAR) and Sum of Pain Intensity Difference(SPID)
Description: The Pain Intensity Difference (PID) at each time point was derived by subtracting the pain intensity from baseline pain intensity, so that a higher value was indicative of a greater improvement. Time weighted SPID for each specified interval (scale ranges from 0 to 10; 0=no pain relief and 10= complete pain relief) was derived by first multiplying each PID score by the time from the previous time point, and adding them together for each scheduled time point within the time interval (e.g., 4-12 hours in case of SPID 4-12). Time weighted TOTPAR for each specified interval was similarly derived.
Time Frame: 0-12 hours after Dose 1
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Time weighted units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Time weighted units on a scale
  TOTPAR 0-12 hours | 54.59 (40.830) | 12.05 (27.114)
  TOTPAR 0-4 hours | 16.84 (11.854) | 3.18 (6.749)
  TOTPAR 4-8 hours | 25.94 (19.013) | 5.34 (12.393)
  TOTPAR 4-12 hours | 43.38 (33.851) | 9.92 (23.411)
  SPID 0-12 hours | 37.20 (34.791) | 0.45 (24.378)
  SPID 0-4 hours | 11.64 (10.222) | -0.18 (6.591)
  SPID 4-8 hours | 17.88 (16.158) | 0.24 (11.034)
  SPID 4-12 hours | 29.49 (28.654) | 0.67 (20.617)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; The PID at each time point prior to dose 2 was derived by substracting the pain intensity from the base line pain intensity, so that a higher value was indicative of a greater improvement. Time weighted SPID for each specified interval was derived by first multiplying each PID score by the time from the previous time point, and adding them together for each scheduled time point within the time interval. Time weighted TOTPAR for ech specified interval was similarly derived; Test type: Superiority or Other; p < 0.0001, ANCOVA; With terms for treatment, gender, and baseline pain score categories stratified as ≤7 and >7

8. Secondary Outcome: Duration of Relief After Dose 1
Description: Duration of relief was defined as the time to treatment failure (i.e.,taking rescue medication, or withdrawing due to lack of efficacy) up to the 12-hour time point. For those withdrawing from the study due to lack of efficacy prior to taking dose 2 or rescue medication, time to treatment failure was the time from dose 1 to the last assesment time. For those discontinuing from the study for any other reason, the time to treatment failure was censored at the last assessment time.
Time Frame: Time to rescue or time of Dose 2 (up to 12 hours following dose 1)
Population: Intention to treat (ITT)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Minutes | 720 [1 to 720] | 101 [1 to 720]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank

9. Secondary Outcome: Percentage of Participants Who Require Rescue Medication at or Prior to Hour 8, Hour 10, and Hour 12 After Taking Dose 1
Description: Percentage of participants who require rescue medication (Lortab) at or prior to hour 8, hour 10 and hour 12 were reported and 95% confidence intervals for the corresponding parameters were calculated.
Time Frame: 0-12 hours after taking Dose 1
Population: Intention to treat (ITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Percentage of participants
  Rescue at or prior to 8 hours after dose 1 | 31.4 [24 to 38] | 82.8 [75 to 91]
  Rescue at or prior to 10 hours after dose 1 | 34.9 [28 to 42] | 85.1 [78 to 93]
  Rescue at or prior to 12 hours after dose 1 | 36.1 [29 to 43] | 85.1 [78 to 93]
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; The proportions of subjects who rescued at or prior to hour 8, hour 10, and hour 12 were reported and 95% confidence intervals for the corresponding parameters were calculated; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

10. Secondary Outcome: Pain Relief and PID Scores at Individual Time Points for Dose 1
Description: Pain relief and pain intensity difference (PID) scores at individual time points were summarized by descriptive statistics. The PID at each time point prior to dose 2 was derived by subtracting the pain intensity from the baseline pain intensity, so that a higher value was indicative of a greater improvement. Range of possible scores could be from 0 (no improvement) to 5 (greatest possible improvement)
Time Frame: 24, 36, 48 hours after taking Dose 1
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale
  24 hours after dose 1. | 3.11 (3.466) | 0.18 (2.599)
  36 hours after dose 1. | 3.10 (3.460) | 0.22 (2.704)
  48 hours after dose 1. | 3.44 (3.756) | 0.22 (2.721)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; The pain relief and PID scores at individual time points were summarized by descriptive statistics. The test and reference were compared at each individual time point at 24, 36 and 48 hours; Test type: Superiority or Other; p < 0.0001, ANCOVA

11. Secondary Outcome: Global Evaluation for Dose 1
Description: Global evaluation for dose 1, either at the time of rescue or at dose 2 (hour 12), whichever came first were summarized. At the 12-hour time point but before Dose 2, or within 1 minute of rescue medication use (if it occurred before hour 12), the subject was to provide a Global Evaluation of Dose 1 of study medication on an 11 point PI-NRS in response to the following command:
  "Select the number that best describes how you would rate this medication as a pain-reliever (select one number only)." The range went from 0 (Very poor) to 10 (Excellent).
Time Frame: At 12 hours after Dose 1 or at time of rescue
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale | 6.05 (3.536) | 1.79 (2.898)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Global evaluation for dose 1, either at the time of rescue or at dose 2 whichever came first were summarized by descriptive statistics based on non-missing data. The range went from 0 (Very poor) to 10 (Excellent) units on an 11-point Pain Intensity Numerical Rating Scale (PI-NRS); Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories

12. Secondary Outcome: Global Evaluation, Maximum Relief, and Overall Relief for Dose 2
Description: Global evaluation, maximum relief, and overall relief scores for dose 2 were summarized with descriptive statistics. The subject was to provide a description for the Global Evaluation, maximum relief and overall relief of Dose 2 of study medication on an 11 point PI-NRS: Global Evaluation: "rate the study medication as a pain-reliever"; Maximum Pain Relief: "maximum pain relief received from the last dose"; Overall Pain Relief: "overall quantity of pain relief received from the last dose". The range went from 0 (Very poor or No relief) to 10 (Excellent or Complete relief).
Time Frame: At 24 hours or at time of rescue between 12 and 24 hours
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale
  Global Evalution for Dose 2 | 6.82 (2.914) | 4.24 (3.673)
  Maximum Relief for Dose 2 | 7.27 (2.997) | 5.02 (3.864)
  Overall Relief for Dose 2 | 6.62 (3.005) | 4.46 (3.588)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Global evaluation scores for dose 2 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide global evaluation of dose 2 study medication using a range that went from 0 (Very poor) to 10 (Excellent) units on an 11-point Pain Intensity Numerical Rating Scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P- value from ANCOVA with terms for treatment, gender and baseline pain score categories
Statistical Analysis 2: Comparison: Ibuprofen 600mg ER vs Placebo; Maximum relief scores for dose 2 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide maximum relief scores for dose 2 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain scores categories
Statistical Analysis 3: Comparison: Ibuprofen 600mg ER vs Placebo; Overall relief scores for dose 2 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide overall relief scores for dose 2 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories

13. Secondary Outcome: Global Evaluation, Maximum Relief, and Overall Relief for Dose 3
Description: Global evaluation, maximum relief, and overall relief scores for dose 3 were summarized with descriptive statistics. The subject was to provide a description for the Global Evaluation, maximum relief and overall relief of Dose 3 of study medication on an 11 point PI-NRS: Global Evaluation: "rate the study medication as a pain-reliever"; Maximum Pain Relief: "maximum pain relief received from the last dose"; Overall Pain Relief: "overall quantity of pain relief received from the last dose". The range went from 0 (Very poor or No relief) to 10 (Excellent or Complete relief).
Time Frame: At 36 hours or at time rescue between 24 and 36 hours
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale
  Global Evaluation for Dose 3 | 7.14 (2.839) | 4.98 (3.549)
  Maximum Relief for Dose 3 | 7.61 (2.922) | 5.63 (3.805)
  Overall Relief for Dose 3 | 6.76 (2.942) | 5.02 (3.634)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Global evaluation scores for dose 3 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide global evaluation of dose 3 study medication using a range that went from 0 (Very poor) to 10 (Excellent) units on an 11-point Pain Intensity Numerical Rating Scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories
Statistical Analysis 2: Comparison: Ibuprofen 600mg ER vs Placebo; Maximum relief scores for dose 3 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide maximum relief of dose 3 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and basee pain score categories
Statistical Analysis 3: Comparison: Ibuprofen 600mg ER vs Placebo; Overall relief scores for dose 3 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide overall relief of dose 3 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories

14. Secondary Outcome: Global Evaluation, Maximum Relief, and Overall Relief for Dose 4
Description: Global evaluation, maximum relief, and overall relief scores for dose 4 were summarized with descriptive statistics. The subject was to provide a description for the Global Evaluation, maximum relief and overall relief of Dose 4 of study medication on an 11 point PI-NRS: Global Evaluation: "rate the study medication as a pain-reliever"; Maximum Pain Relief: "maximum pain relief received from the last dose"; Overall Pain Relief: "overall quantity of pain relief received from the last dose". The range went from 0 (Very poor or No relief) to 10 (Excellent or Complete relief).
Time Frame: At 48 hours or at time of rescue between 36 and 48 hours.
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ibuprofen 600mg ER | Placebo
Number analyzed (Participants) | 169 | 87
Units on a scale
  Global Evalution for Dose 4 | 7.26 (2.953) | 4.70 (3.715)
  Maximum Relief for Dose 4 | 7.66 (2.970) | 5.34 (3.970)
  Overall Relief for Dose 4 | 7.06 (3.045) | 4.89 (3.803)
Statistical Analysis 1: Comparison: Ibuprofen 600mg ER vs Placebo; Global evaluation scores for dose 4 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide global evaluation of dose 4 study medication using a range that went from 0 (Very poor) to 10 (Excellent) units on an 11-point Pain Intensity Numerical Rating Scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories
Statistical Analysis 2: Comparison: Ibuprofen 600mg ER vs Placebo; Maximum relief scores for dose 4 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide maximum relief of dose 4 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories
Statistical Analysis 3: Comparison: Ibuprofen 600mg ER vs Placebo; Overall relief scores for dose 4 were summarized by descriptive statistics. Only non-missing values are used for the summary statistics. The subjects were to provide overall relief of dose 4 study medication on an 11-point pain intensity numerical rating scale (PI-NRS)in response to pain relief; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value from ANCOVA with terms for treatment, gender and baseline pain score categories

ADVERSE EVENTS:
Arm/Group | Ibuprofen 600mg ER | Placebo
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/87
Other Adverse Events (participants affected / at risk) | 0/169 | 0/87

LIMITATIONS AND CAVEATS:
Of the 12 subjects who prematurely discontinued all 4 doses of the study drug, 6 subjects received 1 dose of study drug, 2 subjects received 2 doses, and 4 subjects received 3 doses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less